CLINICAL TRIAL: NCT04201782
Title: Long-Term Follow-up of HIV-Infected Subjects Treated With Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases (SB-728-T or SB-728mR-T)
Brief Title: Long-term Follow-up of HIV Subjects Exposed to SB-728-T or SB-728mR-T
Status: Terminated | Type: Observational
Why Stopped: There have been no significant safety issues in any subjects exposed between 7.5 and 13.5 years ago to either SB-728-T or SB-728mR-T, including no delayed adverse events related to the investigational product.
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: SB-728-1003
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: HIV-1-infection
Keywords: HIV; gene editing; CCR5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — 1. Clinical condition assessment
  2. Chemistry which includes bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), sodium, potassium, chloride, bicarbonate, urea nitrogen, creatinine, total protein, albumin, calcium, and phosphorous.
  3. CBC which includes hemoglobin, hematocrit, platelet count, red cell count, and white cell count with differential count
  4. CD4+ T-cell count
  5. HIV-1 RNA
  6. HIV proviral DNA
  7. Pentamer
  8. Ad5 and SB-728-T immunogenicity
  9. Research blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Long-term follow-up of HIV-infected subjects who received SB-728-T or SB-728mR-T in a previous trial.
  Interventions: Drug: There are no disallowed treatments

INTERVENTIONS:
Drug: There are no disallowed treatments — Genetic: SB-728-T or SB-728mR-T No study drug is administered in this study. Subjects who received SB-728-T or SB-728mR-T in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
Long-term follow-up of HIV-infected subjects who received SB-728-T or SB-728mR-T. Enrolling subjects will be followed for a total of 12 years.

DETAILED DESCRIPTION:
Subjects infected with HIV who have received therapy with SB-728-T or SB-728mR-T will be eligible to participate in this trial. There will be no treatment in this long-term follow-up study. Subjects who choose to enroll into this extension study will be evaluated for a total of 12 years.

ELIGIBILITY:
Inclusion Criteria:

Subjects who have, in previous Sangamo clinical trial received SB-728-T or SB-728mR-T, autologous T-cells genetically modified at the CCR5 gene by zinc finger nucleases and give consent to participate in the long-term follow-up study.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-Infected Subjects who received SB-728-T under BB-IND 14129 or SB-728mR-T under BB-IND 16082.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-03-18 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Long-term safety of treatment with SB-728-T or SB-728mR-T | 12 years
  Number of subjects with SAEs.
  Number of subjects with delayed adverse events associated with administration of SB-728-T or SB-728mR-T, autologous T-cells genetically modified at the CCR5 gene by zinc finger nucleases.
  Incidence of new malignancies, neurologic disorders (new or exacerbation of pre-existing), rheumatologic disease (new or exacerbation of pre-existing), autoimmune disorder (new or pre-existing), and new hematologic disorder.

SECONDARY OUTCOMES:
Long-term effects of SB-728-T or SB-728mR-T on CD4+ T-cell counts and on the viral load and tropism of HIV in blood. | 2 years
  Long-term effects of SB-728-T or SB-728mR-T will be measured by the following:
  CD4+ T-cell counts through Month 24
  HIV co-receptor tropism through Month 24
  Viral load through Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics, Inc.
Locations (4):
- United States (4):
  - Quest Clinical Research, San Francisco, California
  - Circle CARE Center, LLC, Norwalk, Connecticut
  - Orlando Immunology Center, Orlando, Florida
  - Central Texas Clinical Research, Austin, Texas